CLINICAL TRIAL: NCT02641223
Title: Evaluation of Objective Outcomes With the Use of an Activity Tracker During the Trial Period of Spinal Cord Stimulation
Status: Completed | Type: Observational
Sponsor: University of California, Davis (Other)
Responsible Party: Sponsor
Other Study IDs: 7877631
Record Dates: First submitted 2015-12-16; First posted 2015-12-29 (Estimated); Last update posted 2017-05-30 (Actual); Status verified 2017-05

CONDITIONS: Post-laminectomy Syndrome; Axial Back Pain
MeSH Terms: conditions — post laminectomy syndrome

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Device: spinal cord stimulator — Pt asked to wear FitBit device prior to and after spinal cord stimulator placement.

SUMMARY:
For this study the investigators will conduct five-day trial periods for spinal cord stimulator (SCS) effectiveness-once a patient is deemed to be a possible SCS candidate, the trial leads are implanted and they are asked to return to clinic in five days to evaluate the effectiveness of the trial. The primary outcome for this study will be a comparison of daily energy expenditure (EE), in units of kcal/day, prior to and after the trial implantation of the SCS leads and external pulse generator. Patients will wear the accelerometer device twenty-four hours a day for five days prior to the trial lead implantation to obtain baseline values, have the trial leads implanted in the procedure clinic, then continue to wear the accelerometer for another five days. Baseline and post-SCS energy expenditure values will be compared. The secondary outcomes for this study will be steps taken, hours of sleep, and Oswestry Disability Index (ODI, as described in appendix 1) during the pre and post trial implantation periods. SCS itself is not a research procedure in this study, rather it is part of routine medical care for patients who would benefit from the procedure.

ELIGIBILITY:
Inclusion Criteria:

* Patients presenting to the UCD chronic pain clinic with post-laminectomy syndrome and demonstrate signs of neuropathic axial back pain will be considered.

Exclusion Criteria:

* Adults unable to consent, individuals who are not yet adults, pregnant women, patients unable to stop anticoagulation, and prisoners will be excluded.
* Pregnant patients will be excluded due to the risks of radiation exposure during SCS procedures and prisoners will be excluded as our clinic does not receive referrals from prison populations at this time.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Patients presenting to the UCD chronic pain clinic with post-laminectomy syndrome and demonstrate signs of neuropathic axial back pain will be considered. These patients should also be qualified for SCS placement.
Sampling Method: Non-Probability Sample
Enrollment: 9 (Actual)
Dates: Start 2015-11; Primary Completion 2016-12 (Actual); Study Completion 2016-12 (Actual)

PRIMARY OUTCOMES:
Change in daily energy expenditure in units of kcal/day. | 10 days: change in energy expenditure from 5 days prior to SCS implantation and 5 days post SCS implantation.
  Energy expenditure (EE) is measured for five days prior to SCS implantation and the average EE is calculated. After SCS lead implantation, EE is again measured for 5 days and the average EE is calculated. The change in pre and post SCS implantation is examined.

SECONDARY OUTCOMES:
Change in sleep duration in units of minutes. | 10 days: change in sleep duration between 5 days prior to SCS implantation and 5 days post SCS implantation.
  Change in average hours of sleep over a five day period is compared pre and post SCS trial lead implantation.
Change in steps taken in units of number of steps. | 10 days: change in steps taken between 5 days prior to SCS implantation and 5 days post SCS implantation.
  Change in average steps taken over a five day period is compared pre and post SCS trial lead implantation.

CONTACTS AND LOCATIONS:
Locations (1):
- Lawrence J. Ellison Ambulatory Care Center, Sacramento, California, United States